CLINICAL TRIAL: NCT00002275
Title: Lipid-Based Parenteral Nutritional Support in Patients With the Acquired Immunodeficiency Syndrome and Pneumocystis Carinii Pneumonia. A Comparison of Two Lipid Formulations
Brief Title: A Comparison of Two Types of Injected Nutritional Supplements in Patients With AIDS and Pneumocystis Carinii Pneumonia (PCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 041B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Weight Loss; Pneumonia, Pneumocystis carinii; Parenteral Nutrition; Liposyn; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Weight Loss; Pneumonia, Pneumocystis; Hyperphagia; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Drug: Fat Emulsion 2%
Drug: Fat Emulsion 20%

SUMMARY:
The objectives of this study are:

To establish whether there is a difference in clinical effectiveness of Liposyn II 20 percent as compared with Liposyn III 2 percent in AIDS patients with Pneumocystis carinii pneumonia (PCP). To compare the effects of the two lipid emulsions on immunologic function in AIDS patients. To compare the effect of the two lipid emulsions on HIV load in AIDS patients as measured by reverse transcriptase (RT) in culture. To determine whether a decrease in HIV infectivity is greater in patients given a parenteral feeding regimen containing Liposyn II 20 percent or Liposyn III 2 percent.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* All drugs used for the standard treatment of Pneumocystis carinii pneumonia (PCP).
* Other drugs for treatment of other AIDS conditions if they have been started more than 3 months prior to study entry.

Patients must have:

* Diagnosis of AIDS.
* Weight loss > 10 percent of premorbid body weight.
* First or second episode of acute Pneumocystis carinii pneumonia (PCP).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Do Not Resuscitate (DNR) status.
* Biliary stasis.

Patients with the following are excluded:

* Do Not Resuscitate (DNR) status.
* Biliary stasis.

Prior Medication:

Excluded within 3 months of study entry:

* Immunomodulators.
* Antiviral new DT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- East Orange Veterans Administration Med Ctr, East Orange, New Jersey, United States

REFERENCES:
- [Background] Martin DF, Parks DJ, Mellow SD, Ferris FL, Walton RC, Remaley NA, Chew EY, Ashton P, Davis MD, Nussenblatt RB. Treatment of cytomegalovirus retinitis with an intraocular sustained-release ganciclovir implant. A randomized controlled clinical trial. Arch Ophthalmol. 1994 Dec;112(12):1531-9. doi: 10.1001/archopht.1994.01090240037023. PMID 7993207